CLINICAL TRIAL: NCT04644887
Title: The Effect of Dietary Fat Quality Modification for Liver Fat Content in Participants With Different Variants in PNPLA3 Gene - Liver, Diet and Genetic Background (LIDIGE STUDY)
Brief Title: Liver, Diet and Genetic Background
Acronym: LIDIGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LIDIGE
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Liver Fat
Keywords: human; diet; dietary fat; liver fat; genotype; nutrigenomics
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants and investigators are blinded with the genotype, but not with the dietary groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy diet CC genotype (Experimental): The participants will follow the intervention diet during the 12-week intervention period.
  Interventions: Other: Dietary intervention: Healthy diet
- Control diet CC genotype (Active Comparator): The participants will follow the control diet during the 12-week intervention period.
  Interventions: Other: Dietary intervention: Control diet
- Healthy diet GG genotype (Experimental): The participants will follow the intervention diet during the 12-week intervention period.
  Interventions: Other: Dietary intervention: Healthy diet
- Control diet GG genotype (Active Comparator): The participants will follow the control diet during the 12-week intervention period.
  Interventions: Other: Dietary intervention: Control diet

INTERVENTIONS:
Other: Dietary intervention: Healthy diet — Dietary guidance in the intervention group is based on the Nordic and Finnish nutrition recommendations with an emphasis on the quality of dietary fat. The aims for the intake of fatty acids will be SFA < 10 % of energy intake (E%) and mono- and polyunsaturated fatty acids (UFA) >2/3 of the total fat intake. The key food products such as vegetable oil-based spread, liquid margarine and canola oil are provided to the participants. The participants are recommended to use fat free (e.g. milk, sourdough milk and yogurt) and low fat (e.g. cheese ≤ 17%) dairy products and low-fat meat, poultry, and fish as well as natural nuts and seeds.
  Arms: Healthy diet CC genotype; Healthy diet GG genotype
Other: Dietary intervention: Control diet — The control diet corresponds to the average nutrient intake in the Nordic countries, i.e. the intake of SFA about 15 E% and the proportion of UFA about 50 % of total fat intake. The participants of the control group will get butter-based spread for bread and cooking. They are recommended to use semi-skimmed milk (1,5 %), normal fat yogurt (~2%), normal fat cheese (~24-35 %) and avoid consumption of vegetable oils. They are allowed to eat a portion of fish and nuts once a week.
  Arms: Control diet CC genotype; Control diet GG genotype

SUMMARY:
PNPLA3 rs738409 (I148M) variant is associated with hepatic liver accumulation and chronic liver diseases including non-alcoholic fatty liver disease. It has been shown that obesity augments genetic risk but studies investigating the interaction of PNPLA3 rs738409 risk variant and diet are scarce. The aim is to investigate the effect of dietary fat quality modification in participants with different variants of the PNPLA3 gene (rs738409). The primary outcome is the change in liver fat measured by magnetic resonance imaging in the randomized controlled 12-week dietary intervention trial.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common liver disease worldwide. The composition of the diet, especially quality of dietary fat, contributes to the susceptibility to hepatic lipid accumulation. Saturated fatty acids (SFA), but not polyunsaturated fatty acids (PUFA) increases intrahepatic triglycerides with and without concomitant weight gain. Therefore, the modification of dietary fat quality is the key dietary approach for the prevention of NAFLD.

PNPLA3 rs738409 (I148M) variant is associated with hepatic liver accumulation and chronic liver diseases including NAFLD. It has been shown that obesity augments genetic risk but studies investigating the interaction of PNPLA3 rs738409 risk variant and diet are scarce. Therefore, the aim is to investigate the effect of dietary fat quality modification (high unsaturated fat vs. high SFA) on liver fat and lipid and glucose metabolism in participants with different variants (CC or GG) of the PNPLA3 gene.

The investigators will conduct the randomized controlled 12-week dietary intervention trial in participants with different homozygous PNPLA3 variants (CC or GG). The primary outcome of the intervention is in the amount of liver fat measured by nuclear magnetic resonance imaging (MRI). Altogether 140 homozygous participants (PNPLA3 rs738409 CC and GG) will be recruited from the Metabolic Syndrome in Men (METSIM) study. The inclusion criteria include BMI < 35 kg/m2 and age < 75 years. The main exclusion criteria include diabetes, acute illness, or current evidence of acute or chronic inflammatory or infective diseases.

Dietary guidance in the intervention group is based on the Nordic and Finnish nutrition recommendations with an emphasis on the quality of dietary fat. The aims for the intake of fatty acids will be SFA < 10 % of energy intake (E%) and mono- and polyunsaturated fatty acids (UFA) >2/3 of the total fat intake.

The diet of the control group corresponds to the average nutrient intake in the Nordic countries, i.e. the intake of SFA about 15 E% and the proportion of UFA about 50 % of total fat intake.

ELIGIBILITY:
Inclusion Criteria:

* PNPLA3 rs738409, CC or GG
* Body mass index (BMI) < 35 kg/m2
* Total cholesterol < 8 mmol/l
* LDL cholesterol < 5 mmol/l
* Fasting plasma glucose < 7 mmol/l
* Plasma alanine aminotransferase (ALT) < 100 U/l
* Age 60-75 y

Exclusion Criteria:

The main exclusion criteria include acute illness or current evidence of acute or chronic inflammatory or infective diseases. No patients with hepatitis B and/or C, autoimmune hepatitis, Wilsons disease/alpha-1-antitrypsin deficiency, hemochromatosis, chronic kidney disease, unstable hypothyroidism or lipoatrophy will be accepted. No subjects with diagnosed diabetes (any type) are accepted. In addition to that, no diagnosed depression or any mental illness rendering the patients unable to understand the nature, scope and possible sequences of the study will be accepted. Alcohol abuse (daily consumption ≥ 30 g for men and ≥ 20 g for women) is also exclusion criteria.

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men because the population source for recruitment Metabolic syndrome in men (METSIM) study is composed solely by men.
Enrollment: 99 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Liver fat | 12 weeks
  The primary outcome is the change in liver fat measured by magnetic resonance imaging

SECONDARY OUTCOMES:
Hepatic condition monitored by ultrasound | 12 weeks
  The hepatic condition will be monitored by ultrasound
Hepatic condition monitored by elastography | 12 weeks
  The hepatic condition will be monitored by elastography
Hepatic condition monitored by calculated indexes | 12 weeks
  The hepatic condition will be monitored by calculating and comparing Fibrosis-4 index, NAFLD Fibrosis Score, hepatic steatosis index, the fatty liver index and NAFLD liver fat score.
Glucose metabolism | 12 weeks
  Changes in glucose metabolism (oral glucose tolerance test, 0, 30 min and 2 h samples)
Serum lipid profile | 12 weeks
  Concentrations of total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides
Inflammatory markers | 12 weeks
  Serum circulating concentrations of high-sensitivity C-reactive protein
Plasma metabolomic profile | 12 weeks
  Mass spectrometry based metabolomics analysis
Plasma lipidomic profile | 12 weeks
  Mass spectrometry based lipidomics analysis
Gut microbiota | 12 weeks
  The DNA/RNA of gut microbiota will be extracted and collected for high throughput metagenomics and metatranscriptomics to observe changes in type and composition of gut microbiota.
Fatty acid composition of plasma lipid fractions | 12 weeks
  Fatty acid composition of plasma phospholipids, cholesteryl esters and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schwab, Professor, Principal Investigator — University of Eastern Finland
Locations (1):
- Institute of Public Health and Clinical Nutriton, Kuopio, Finland